CLINICAL TRIAL: NCT06877039
Title: Observational Study on the Characteristics of Clinical Laboratory Indicators in Patients with Dengue Fever
Brief Title: Characteristics of Clinical Laboratory Indicators in Patients with Dengue Fever
Status: Completed | Type: Observational
Sponsor: Foshan Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Qilong Nie, Director, Foshan Hospital of Traditional Chinese Medicine
Other Study IDs: Foshan Hospital of Traditional
Record Dates: First submitted 2025-02-27; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational studies did not involve any interventions

SUMMARY:
The objective of this observational study was to understand the changes in laboratory indicators and clinical manifestations of dengue patients at various ages, and to provide new ideas for the treatment and prevention of dengue. The main questions it aims to answer are: 1 What are the key abnormal items in blood routine indicators of dengue patients? 2 Does dengue affect liver function in patients? Will there be liver damage? And when? 3. What are the specific clinical manifestations of dengue patients?

ELIGIBILITY:
* Inclusion Criteria**:

  * Meet the clinical diagnostic criteria for dengue fever, with blood indicators showing that the dengue antigen is positive.
  * No age limit for inclusion.
  * Voluntarily agree to participate in the study and sign the informed consent.
  * Complete clinical data available, including symptoms and laboratory tests, to support subsequent analysis.
* Exclusion Criteria**:

  * Incomplete or unavailable clinical data. Patients will be excluded if sufficient laboratory data and symptoms cannot be collected.
  * Unable to understand or unwilling to sign the informed consent for any reason.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects in this study were dengue fever patients.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
WBC | From January 2024 to December 2024
  WBC (White Blood Cell count), unit: cells/µL. All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
HGB (Hemoglobin) | From January 2024 to December 2024
  HGB (Hemoglobin), unit: g/dL; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
PLT (Platelet count) | From January 2024 to December 2024
  PLT (Platelet count), unit: cells/µL; All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.
ANC (Absolute Neutrophil Count) | From January 2024 to December 2024
  ANC (Absolute Neutrophil Count), unit: cells/µL. All these markers will be assessed at baseline (Day 0) and during monthly follow-up visits throughout the study period from January 2024 to December 2024. Data will be collected and summarized as.

CONTACTS AND LOCATIONS:
Locations (1):
- Foshan Hospital of Traditional Chinese Medicine, Guangzhou University of Chinese Medicine, Foshan, 528051, Guangdong, China., Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No